CLINICAL TRIAL: NCT00744289
Title: A Randomised Controlled Trial to Evaluate the Effectiveness of a Small Financial Incentive After the Second and Third Dose of a Hepatitis B Vaccine, on Vaccine Completion in People Who Inject Drugs
Brief Title: Hepatitis B Acceptability and Vaccination Incentive Trial
Acronym: HAVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Professor Lisa Maher, The Kirby Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: X08-0161
Record Dates: First submitted 2008-08-26; First posted 2008-08-29 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; People who inject drugs; Financial incentive; Vaccine completion
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (No Intervention): Participants in Arm 1 will not receive any financial incentive after the second and third dose of hepatitis B vaccine have been administered.
- Arm 2 (Other): Participants in Arm 2 will receive a small financial incentive after the second and third dose of the hepatitis B vaccine
  Interventions: Other: Incentive condition

INTERVENTIONS:
Other: Incentive condition — Receipt of a small financial incentive after the second and third dose of the hepatitis B vaccine
  Arms: Arm 2

SUMMARY:
Aims:

This prospective trial seeks to investigate the efficacy of a financial incentive in increasing the uptake and completion of the HBV vaccine series among people who inject drugs (PWID). Using a randomised controlled trial design, the investigators will offer the 3 dose, accelerated HBV schedule to eligible PWID allocated to either a standard of care or incentive condition. Participants allocated to the incentive condition will receive a small incentive payment after the second and third dose of the vaccine. It is hypothesized that the proportion of participants who complete the vaccine series in the incentive payment arm will be higher compared to the non-incentive payment arm (standard of care).

DETAILED DESCRIPTION:
Injecting drug use is the leading exposure category for notifications of newly acquired hepatitis B virus (HBV) infection in Australia. Despite the existence of a safe and efficacious vaccine, hepatitis B coverage remains low among Australian people who inject drugs (PWID) and little is known about attitudes to immunisation, barriers to uptake and willingness to participate in vaccine trials among this group. Candidate vaccines for hepatitis C virus (HCV) and HIV are currently in development and HBV immunisation provides a surrogate for examining strategies to deliver vaccines to this group.

Secondary objectives of this trial are to (i) assess the cost effectiveness of the interventions; (ii) identify the correlates of immunity in this group; (iii) assess the acceptability of vaccines, including HBV vaccines, barriers to immunisation uptake and willingness to participate in vaccine trials among PWID; and (iv) assess hepatitis B-related knowledge in this group.

Research Design: A total of 200 eligible PWID or people at risk of initiating injecting (those with no history of exposure to or receipt of more than one vaccination against HBV) will be recruited and interviewed prior to randomisation on a 1:1 basis (100 per arm) to either the (1) control (standard of care) or (2) incentive conditions. All participants will be offered the 3 dose accelerated vaccine schedule (20ug at 0, 7 and 21 days) and will be followed up at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years and above.
* Injected drugs at least once in the preceding six months, OR (i) Use of any illegal/non-prescription drug apart from cannabis (e.g., speed, coke, ice, heroin) in the last three months, AND (ii) Spent time with 2 or more people who inject drugs on a weekly or more frequent basis in the last three months.
* No previous hepatitis B infection, and a maximum of one previous dose of hepatitis B vaccination, or unknown infection and vaccination status, based on self-report and, where available, medical records
* Ability to provide informed consent, to be randomized and attend vaccinations over a period of three weeks and to attend follow-up at 12 weeks post-randomisation.

Exclusion Criteria:

* Evidence of natural or vaccine-induced immunity.
* Previous exposure or two+ vaccinations (as identified by self-report), where HBV surface antibody >= 10 mIU/ml
* Serious mental or physical illness or disability likely to impact on capacity to complete the study procedures
* Insufficient English language skills that will impair ability to give informed consent or provide reliable responses to study interviews /questionnaires
* Human Immunodeficiency Virus infection
* Refusal to be vaccinated against Hepatitis B Virus (HBV)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Determine, relative to a 'standard of care' control condition, the efficacy of incentive payments to increase HBV vaccine completion using an accelerated schedule (0, 7, and 21 days). | 12 weeks

SECONDARY OUTCOMES:
Assess the relative cost effectiveness of standard care compared to incentive payments as methods of improving rates of successful vaccine series completion and vaccine-induced immunity | 12 weeks
Identify the correlates of immunity (defined as hepatitis B surface antibody levels greater than 10 mIU/ml) | At baseline and week 12
Assess the acceptability of vaccines, including HBV vaccines, barriers to immunisation uptake and willingness to participate in vaccine trials among PWID | At baseline and week 12
Assess hepatitis B-related knowledge in this group | At baseline and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Maher, PhD, Principal Investigator — Kirby Institute
Locations (1):
- The Kirby Institute, Sydney, New South Wales, Australia